CLINICAL TRIAL: NCT05619718
Title: Loneliness Group Intervention for Geriatric Psychiatry Inpatients
Brief Title: Loneliness Group Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12528
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Loneliness
Keywords: loneliness; geriatric; functional analytic psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group will receive Awareness, Courage, and Love Groups for loneliness.
  Interventions: Behavioral: Awareness, Courage, and Love Groups
- Control (Active Comparator): Control group will receive treatment as usual in the form of Mutual Help Meetings.
  Interventions: Other: Mutual Help Meetings

INTERVENTIONS:
Behavioral: Awareness, Courage, and Love Groups — Groups based on the Awareness, Courage, and Love framework from functional analytic psychotherapy
  Arms: Treatment
Other: Mutual Help Meetings — Groups based on treatment as usual where patients gather to discuss how they can help others on the ward, and make requests for how others can help them.
  Arms: Control

SUMMARY:
The goal of this pilot study is to determine the feasibility and acceptability of a group loneliness intervention in geriatric psychiatry inpatients. This type of group loneliness intervention is based on functional analytic psychotherapy and is called Awareness, Courage, and Love Groups.

DETAILED DESCRIPTION:
The objective of our clinical trial is to adapt, implement, and evaluate a type of loneliness group intervention called Awareness, Courage, and Love Groups for older adults in a psychiatric unit. The following research questions will be answered: (a) Are ACL groups with geriatric psychiatry inpatients feasible and acceptable? (b) Do such ACL groups demonstrate preliminary efficacy?

ELIGIBILITY:
Inclusion Criteria:

* Admission to geriatric psychiatry inpatient unit

Exclusion Criteria:

* Individuals who are disoriented to person, delirious, unable to tolerate or participate meaningfully in the group, or otherwise unable to provide consent to research and psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2027-08-25 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Inclusion of Other in the Self Scale (IOS) | Up to 2 months
  Brief single-item pictorial measure of social closeness. The minimum value is 1, the maximum value is 7, and higher scores indicate a better outcome.
UCLA Loneliness Scale (ULS-6) | Up to 2 months
  Brief measure of loneliness. The minimum value is 6, the maximum value is 24, and higher scores indicate a worse outcome.
Relational Health Indices (RHI) | Up to 2 months
  Brief measure of group relational health. The minimum value is 8, the maximum value is 40, and higher scores indicate a better outcome.
Quantitative Program Satisfaction | Up to 2 months
  Brief measure of program satisfaction. The minimum value is 0, the maximum value is 16, and higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Cantril Self-Anchoring Striving Scale | Up to 2 months
  1 item pictorial scale of subjective wellbeing from 0 (minimum) to 10 (maximum). A higher score indicates a better outcome.
Sacred Moment Qualities (SMQ) | Up to 2 months
  Brief measure of perceived sacred qualities, adapted from Pargament et al. (2014). The minimum value is 11, the maximum value is 55, and higher scores indicate a better outcome.

OTHER OUTCOMES:
Satisfaction Questionnaire | Up to 2 months
  Brief open-ended questions about program satisfaction. Responses are qualitative.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth VanBussel, MD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- Parkwood Institute Mental Health, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT05619718/Prot_SAP_000.pdf